CLINICAL TRIAL: NCT00046436
Title: Mother-Infant Rapid Intervention at Delivery (MIRIAD)
Brief Title: Rapid HIV Tests for Women Late in Pregnancy and During Labor
Status: Terminated | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Other Study IDs: PACTG P1031
Record Dates: First submitted 2002-09-30; First posted 2002-10-01 (Estimated); Last update posted 2013-06-03 (Estimated); Status verified 2013-05

CONDITIONS: HIV Infections
Keywords: AIDS Serodiagnosis; Pregnancy Complications, Infectious; Anti-HIV Agents; Disease Transmission, Vertical
MeSH Terms: conditions — HIV Infections; Pregnancy Complications, Infectious

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study will look at how well the OraQuick HIV 1/2 Antibody rapid test works and how women accept being tested for HIV late in pregnancy and during labor. For women with positive test results, the study will look at whether or not these women accept anti-HIV drugs and which drugs they receive.

DETAILED DESCRIPTION:
A simple HIV test design and easily interpretable, fast results are logistical advantages in clinical settings such as the labor and delivery unit. A fast test result means that a woman can make important choices about her and her baby's medical care before she delivers her baby. If a woman finds out she has HIV, she can decide to take antiretroviral drugs before delivery to decrease the risk of passing HIV to her baby. These advantages are also important for women with little or no prenatal care who present for care late in pregnancy, but may not be inclined to return for a standard test result or adhere to subsequent prenatal visits.

Eligible women who elect to participate in this study will be enrolled in either the Late Presenter Group (women who are not in active labor, and for whom delivery is not imminent) or the Peripartum Group (women who are in active labor with anticipation of delivery within 24 hours). Step I for all women will include rapid HIV testing with OraQuick HIV 1/2 and standard testing with enzyme-linked immunosorbant assay (EIA) or Western blot. Women with a positive HIV test and their infants will be offered preventative antiretroviral therapy and enrollment into Step II. Step II will include clinical evaluations, laboratory evaluations, and an adherence assessment for the women and their infants. Women in the Late Presenter Group who participate in Step II will have one prenatal visit, a visit at labor and delivery, and three postpartum visits. Women in the Peripartum Group who participate in Step II will have three postpartum visits. All infants in Step II will have five study visits through 24 weeks of age.

All antiretroviral drugs will be obtained by prescription and will not be provided through this study.

ELIGIBILITY:
INCLUSION CRITERIA

Late Presenter Group:

* Unknown HIV serostatus
* >= 34 weeks gestation

Peripartum Group:

* Unknown HIV serostatus
* >= 24 weeks gestation
* In active labor or delivery expected within 24 hours

Infants:

* Maternal Step I enrollment
* Positive maternal OraQuick and/or EIA/Western blot result

EXCLUSION CRITERIA

Late Presenter Group:

* Previous or current antiretroviral therapy for treatment of HIV infection
* In active labor
* Evidence of ruptured membranes

Peripartum Group:

* Previous or current antiretroviral therapy for treatment of HIV infection

Min Age: 13 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 7500
Dates: Study Completion 2004-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Maupin, Jr., MD, Study Chair — Louisiana State University Health Sciences Center in New Orleans
Locations (1):
- Univ. of Pennsylvania Health System, Hosp. of the Univ. of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Minkoff H, O'Sullivan MJ. The case for rapid HIV testing during labor. JAMA. 1998 Jun 3;279(21):1743-4. doi: 10.1001/jama.279.21.1743. No abstract available. PMID 9624029
- [Background] Kelen GD, Shahan JB, Quinn TC. Emergency department-based HIV screening and counseling: experience with rapid and standard serologic testing. Ann Emerg Med. 1999 Feb;33(2):147-55. doi: 10.1016/s0196-0644(99)70387-2. PMID 9922409
- [Background] Guay LA, Musoke P, Fleming T, Bagenda D, Allen M, Nakabiito C, Sherman J, Bakaki P, Ducar C, Deseyve M, Emel L, Mirochnick M, Fowler MG, Mofenson L, Miotti P, Dransfield K, Bray D, Mmiro F, Jackson JB. Intrapartum and neonatal single-dose nevirapine compared with zidovudine for prevention of mother-to-child transmission of HIV-1 in Kampala, Uganda: HIVNET 012 randomised trial. Lancet. 1999 Sep 4;354(9181):795-802. doi: 10.1016/S0140-6736(99)80008-7. PMID 10485720
- [Background] Shaffer N, Chuachoowong R, Mock PA, Bhadrakom C, Siriwasin W, Young NL, Chotpitayasunondh T, Chearskul S, Roongpisuthipong A, Chinayon P, Karon J, Mastro TD, Simonds RJ. Short-course zidovudine for perinatal HIV-1 transmission in Bangkok, Thailand: a randomised controlled trial. Bangkok Collaborative Perinatal HIV Transmission Study Group. Lancet. 1999 Mar 6;353(9155):773-80. doi: 10.1016/s0140-6736(98)10411-7. PMID 10459957
- [Background] Bulterys M, Jamieson DJ, O'Sullivan MJ, Cohen MH, Maupin R, Nesheim S, Webber MP, Van Dyke R, Wiener J, Branson BM; Mother-Infant Rapid Intervention At Delivery (MIRIAD) Study Group. Rapid HIV-1 testing during labor: a multicenter study. JAMA. 2004 Jul 14;292(2):219-23. doi: 10.1001/jama.292.2.219. PMID 15249571
- [Background] Jamieson DJ, O'Sullivan MJ, Maupin R, Cohen M, Webber MP, Nesheim S, Lampe M, Garcia P, Lindsay M, Bulterys M. The challenges of informed consent for rapid HIV testing in labor. J Womens Health (Larchmt). 2003 Nov;12(9):889-95. doi: 10.1089/154099903770948113. PMID 14670168